CLINICAL TRIAL: NCT03399695
Title: Comparison of Efficacy and Tolerance of Preoxygenation Using High Flow Oxygen and Face Mask Breathing in Healthy Volunteers.
Brief Title: Preoxygenation Using High Flow Oxygen : Efficacy and Tolerance in Healthy Volunteers
Acronym: PreOx-OHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID RCB 2017-A02343-50
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia; Airway Morbidity; Safety Issues
Keywords: preoxygenation; high flow oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): spontaneous breathing through a face mask connected to the anaesthesia machine delivering 100% oxygen gas flow (15l/min)
  Interventions: Procedure: preoxygenation
- ohd (Experimental): spontaneous breathing through a nasal cannula connected to an humidifier device delivering warm (37°C) high flow oxygen(60l/min)
  Interventions: Procedure: preoxygenation

INTERVENTIONS:
Procedure: preoxygenation — spontaneous breathing

SUMMARY:
High flow nasal cannula oxygen has been proposed to perform preoxygenation in patients with acute respiratory failure requiring orotracheal intubation in intensive care units. However, its use for preoxygenation before the induction of general anaesthesia in operating room has never been evaluated in term of end tidal oxygen fraction which is the gold standard measurement during preoxygenation before general anaesthesia.

The goal of the present study is to measure end tidal oxygen after 3 min of preoxygenation using the recommended method (spontaneous breathing of 100% inhaled oxygen through a face mask) and using high flow nasal canula oxygen, in healthy volunteers.

DETAILED DESCRIPTION:
High flow nasal cannula oxygen has been proposed to perform preoxygenation in patients with acute respiratory failure requiring orotracheal intubation in intensive care units. The results suggest that high flow oxygen could be superior to bag reservoir face mask in term of occurrence of severe hypoxemia during the intubation procedure.

At the present time its use for preoxygenation before the induction of general anaesthesia in operating room has never been evaluated in term of end tidal oxygen fraction which is the gold standard measurement ensuring that the functional residual capacity has been filled with oxygen.

We planned a randomised cross over study in healthy volunteers studying efficacy and tolerance of preoxygenation using spontaneous ventilation with 100% inhaled oxygen through a face mask connected to the anaesthesia machine and preoxygenation using high flow nasal cannula oxygen (60l/min).

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers,
* signed contentment

Exclusion Criteria:

* any chronic or acute disease,
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
FeO2 at 3 min | 3 minutes
  end tidal oxygen fraction measured through a gas analyser

SECONDARY OUTCOMES:
time to obtain an FeO2 at 90% | 6 minutes
  time to obtain an end tidal oxygen fraction measured at 90% measured through a gas analyser
proportion of adequate preoxygenation at 3 min | 6 minutes
  proportion of adequate preoxygenation (FeO2=90%) at 3 min
tolerance | 1 hour
  self reported tolerance on a likert scale
tolerance on VAS | 1 hour
  self reported tolerance on a visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanouz JL, Lhermitte D, Gerard JL, Fischer MO. Comparison of pre-oxygenation using spontaneous breathing through face mask and high-flow nasal oxygen: A randomised controlled crossover study in healthy volunteers. Eur J Anaesthesiol. 2019 May;36(5):335-341. doi: 10.1097/EJA.0000000000000954. PMID 30664524